CLINICAL TRIAL: NCT03830177
Title: Safety and Efficacy of a Topical Scalp Treatment for Dry Scalp Conditions in Children and Adults
Brief Title: Safety and Efficacy of a Topical Scalp Treatment for Dry Scalp Conditions in Children and Adult
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-2309
Record Dates: First submitted 2018-11-27; First posted 2019-02-05 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Dermatitis, Seborrheic; Dry Skin; Eczema
MeSH Terms: conditions — Dermatitis, Seborrheic; Eczema

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): All participants receive a topical scalp treatment containing Lactobacillus sp., honey, and turmeric. Adults apply the treatment daily for 14 days, while children apply it 2-3 times weekly for 14 days.
  Interventions: Drug: Natural Treatment

INTERVENTIONS:
Drug: Natural Treatment — Participants will receive a topical treatment formulated with natural ingredients (Lactobacillus sp., honey, and turmeric) and a kit containing all necessary materials, including an instruction handout. The treatment is applied to the scalp, left for roughly 5 minutes, and rinsed off.
  Other Names: Yobee

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel topical treatment for dry scalp conditions, including dandruff, seborrheic dermatitis, and atopic dermatitis. The study investigates clinical improvements in symptom severity, participant experience with the treatment, and changes in the scalp microbiome before and after use. By studying this treatment, the investigators aim to provide children and adults with a natural, effective option for managing dry scalp conditions.

DETAILED DESCRIPTION:
This study evaluates the safety and efficacy of a novel topical scalp treatment for dry scalp conditions, including dandruff, seborrheic dermatitis, and atopic dermatitis. The treatment contains Lactobacillus sp., honey, and turmeric in an emollient base, hypothesized to alleviate symptoms by addressing microbial imbalances, reducing inflammation, and promoting scalp hydration.

The study will enroll 15-40 pediatric participants aged 1-17 years and 20-40 adults aged 18 and older, all clinically diagnosed with dry scalp. All participants will apply the treatment over a 14-day period. Adults will use the treatment daily, while pediatric participants will apply it 2-3 times weekly. Other scalp therapies will be discontinued during the study period.

The study aims to explore the treatment's potential to improve clinical severity, enhance quality of life, and positively impact the scalp microbiome, providing a natural, effective option for managing dry scalp conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 year (or corrected age of 1 year, for those born prematurely) to 17 years for children, and adults 18 and older
2. Patients with dry scalp and dandruff symptoms as determined by a board-certified Dermatologist, Allergist, or Pediatrician
3. Good general health
4. Participant and/or their parents are able to read, write, and understand study materials in English

Exclusion Criteria:

1. Infants younger than 1 year old
2. Patients diagnosed with other scalp diseases such as psoriasis, tinea capitis, and pediculosis capitis
3. Systemic steroid or oral antibiotic use during the past two months
4. Allergy to any of the preparation components

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Bilaver, PHD, Principal Investigator — Feinberg School of Medicine- Northwestern
Locations (1):
- Medical Dermatology Associates of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol initially planned for 80 participants, but 77 were successfully enrolled at baseline across the two groups - child and adult.
Groups:
- Intervention Arm: The intervention arm includes two subgroups - adults and children. All participants receive a topical scalp treatment containing Lactobacillus sp., honey, and turmeric. Adults apply the treatment daily for 14 days, while children apply it 2-3 times weekly for 14 days.
Period: Overall Study
Arm/Group | Intervention Arm
Started | 77
Adult | 35
Child | 42
Completed | 77
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: All participants receive the topical scalp treatment containing Lactobacillus, honey, and turmeric. Adult participants apply the treatment daily for 14 days, while child participants apply the treatment 2-3 times weekly for 14 days. This arm contains two subgroups for analysis - children and adults.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed in the row refers specifically to the subgroup in the row title. 35 adult samples were analyzed. 42 child samples were analyzed. Combined, 77 samples were analyzed.
  Participants
    Adults: number analyzed (Participants) | 35
    Adults: <=18 years | 0
    Adults: Between 18 and 65 years | 35
    Adults: >=65 years | 0
    Children: number analyzed (Participants) | 42
    Children: <=18 years | 42
    Children: Between 18 and 65 years | 0
    Children: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in the row refers specifically to the subgroup in the row title. 35 adult samples were analyzed. 42 child samples were analyzed. Combined, 77 samples were analyzed.
  Participants
    Adults: number analyzed (Participants) | 35
    Adults: Female | 19
    Adults: Male | 16
    Children: number analyzed (Participants) | 42
    Children: Female | 27
    Children: Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in the row refers specifically to the subgroup in the row title. 35 adult samples were analyzed. 42 child samples were analyzed. Combined, 77 samples were analyzed.
  Participants
    Adults: number analyzed (Participants) | 35
    Adults: American Indian or Alaska Native | 0
    Adults: Asian | 17
    Adults: Native Hawaiian or Other Pacific Islander | 0
    Adults: Black or African American | 2
    Adults: White | 14
    Adults: More than one race | 2
    Adults: Unknown or Not Reported | 0
    Children: number analyzed (Participants) | 42
    Children: American Indian or Alaska Native | 0
    Children: Asian | 3
    Children: Native Hawaiian or Other Pacific Islander | 0
    Children: Black or African American | 2
    Children: White | 20
    Children: More than one race | 11
    Children: Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Determined Using the Investigator's Global Assessment (IGA) - Adult
Description: The Investigator's Global Assessment (IGA) is a 5-point scale used to evaluate the severity of dry scalp conditions. Scores range from 0 (clear) to 4 (severe disease), based on clinical signs such as flaking, erythema, and pruritus. Assessments were conducted at baseline and endpoint to evaluate the efficacy of the treatment in reducing symptom severity.
Time Frame: Baseline, 2 weeks (Study Endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Arm: All participants receive the topical scalp treatment containing Lactobacillus, honey, and turmeric. Adult participants apply the treatment daily for 14 days.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 35
units on a scale
  Baseline | 2.1 (0.6)
  Endpoint | 1.1 (0.8)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p < 0.001, t-test, 1 sided

2. Primary Outcome: Efficacy Determined Using the Investigator's Global Assessment (IGA) - Child
Description: as for outcome 1
Time Frame: Baseline, 2 weeks (Study Endpoint)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention Arm: All participants receive the topical scalp treatment containing Lactobacillus, honey, and turmeric. Child participants apply the treatment 2-3 times weekly for 14 days.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 42
units on a scale
  Baseline | 3.0 [2.8 to 3.3]
  Endpoint | 2.0 [1.8 to 2.2]
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p < 0.001, t-test, 1 sided

3. Primary Outcome: Efficacy Determined Using the Total Severity Scale (TSS) - Adult
Description: The Total Severity Scale (TSS) evaluates the severity of dry scalp conditions by averaging individual scores for erythema, scaling, and pruritus of scalp lesions. Each component is scored on a 4-point scale, ranging from 0 (none) to 3 (severe). The TSS is calculated by summing the scores of individual subscales, each representing a key symptom or feature of the condition, for a total possible score range of 0 to 9, with higher scores indicating greater severity. TSS assessments were conducted at baseline and 2 weeks (Study Endpoint) to determine the treatment's efficacy in reducing symptom severity.
Time Frame: Baseline, 2 weeks (Study Endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 35
units on a scale
  Baseline | 3.5 (1.4)
  Endpoint | 1.8 (1.0)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p < 0.001, t-test, 1 sided

4. Primary Outcome: Efficacy Determined Using the Total Severity Scale (TSS) - Child
Description: as for outcome 3
Time Frame: Baseline, 2 weeks (Study Endpoint)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 42
units on a scale
  Baseline | 3.6 [3.1 to 4.2]
  Endpoint | 1.8 [1.3 to 2.2]
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p < 0.001, t-test, 1 sided

5. Secondary Outcome: Change in Bacterial Composition of Scalp Using RODAC
Description: This exploratory outcome assesses whether the topical treatment alters the scalp microbiome to more closely resemble that of a healthy scalp. Scalp samples were collected at baseline and endpoint using swabs and analyzed with 16S ribosomal RNA (rRNA) sequencing for bacterial diversity and internal transcribed spacer (ITS) sequencing for fungal diversity. Colony counts were measured using the Replicate Organism Detection and Counting (RODAC) method to evaluate bacterial and fungal load changes.
Time Frame: 6 months
Population: Although microbiome samples were collected, no laboratory analysis was conducted, and no data were generated for this outcome measure. As a result, there are no available results to report. There is absolutely no possibility of future analysis.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life Change - Adult
Description: Quality of life was assessed using the ScalpDex-23, a validated 23-item instrument designed to evaluate the impact of scalp dermatitis on symptoms, functioning, and emotions. Each item is scored on a 5-point Likert-type scale ('Never' = 0, 'Rarely' = 25, 'Sometimes' = 50, 'Often' = 75, 'All the time' = 100), with higher scores indicating greater impairment. Subscale scores were calculated for Symptoms (7 items), Emotion (8 items), and Functioning (8 items) by averaging the respective item scores. The total ScalpDex-23 score was calculated as the average of the three subscale scores, yielding a final value ranging from 0 to 100. Assessments were conducted at Baseline and after 2 weeks (Study Endpoint) to measure changes over time.
Time Frame: Baseline, 2 weeks (Study Endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 35
units on a scale
  Baseline | 46 (13.4)
  Endpoint | 39.5 (10.3)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p < 0.001, t-test, 1 sided

7. Secondary Outcome: Quality of Life Change - Child
Description: Quality of life was assessed using the ScalpDex-23, a validated 23-item instrument designed to evaluate the impact of scalp dermatitis on symptoms, functioning, and emotions. Each item is scored on a 5-point Likert-type scale ('Never' = 0, 'Rarely' = 25, 'Sometimes' = 50, 'Often' = 75, 'All the time' = 100), with higher scores indicating greater impairment. Subscale scores were calculated for Symptoms (7 items), Emotion (8 items), and Functioning (8 items) by averaging the respective item scores. The total ScalpDex-23 score was calculated as the average of the three subscale scores, yielding a final value ranging from 0 to 100. Originally, assessments were to be conducted at baseline and endpoint to measure changes in quality of life. However, for children, only midpoint data were collected, so change could not be measured.
Time Frame: 1 week (Study midpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 42
units on a scale | 44.2 (21.1)

ADVERSE EVENTS:
Time Frame: Data was collected over the course of 14 days. Not all participants began the study on the same day.
Description: No difference in definitions.
Groups:
- Adults: All adults in the study will receive the treatment for dry scalp.
  Natural Treatment: The participant will be given the treatment, which contains all natural ingredients, and a kit of all necessary materials to take home with them, which will include a set of instructions. The kit will contain the instruction handout and their treatment. They will be instructed to apply the treatment to their scalp, wait seven minutes, and then rinse their scalp. They will perform this entire procedure once per day for 14 days.
- Children: All children in the study will receive the treatment for dry scalp.
  Natural Treatment: The participant will be given the treatment, which contains all natural ingredients, and a kit of all necessary materials to take home with them, which will include a set of instructions. The kit will contain the instruction handout and their treatment. They will be instructed to apply the treatment to their scalp, wait seven minutes, and then rinse their scalp. They will perform this entire procedure once per day for 14 days.
Arm/Group | Adults | Children
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/42
Other Adverse Events (participants affected / at risk) | 0/35 | 0/42

LIMITATIONS AND CAVEATS:
RODAC: Though scalp swabs were collected, no microbiome data were generated as analysis did not occur. Due to budgetary constraints, RODAC plate analysis was not conducted. The study is now closed, and the IRB is being finalized. Thus, no data are available for this outcome. There is no possibility of future analysis.

Child SCALPDEX: Statistical analysis could not be performed since endpoint data were not collected. Thus, changes in quality of life for this subgroup could not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03830177/Prot_SAP_000.pdf